CLINICAL TRIAL: NCT00344253
Title: A Monocentric, Randomized, Controlled Trial to Test the Efficacy of Interferon-beta in the Treatment of Disseminated Encephalomyelitis (ED)-Associated and Primary Intermediate Uveitis in Comparison to Standard Treatment (TEAM)
Brief Title: Randomized, Controlled Trial to Test the Efficacy of Interferon Beta in the Treatment of Intermediate Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Serono GmbH (Unknown)
Responsible Party: Principal Investigator, Friederike Mackensen, PD Dr. med., Heidelberg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT-Number: 2004-004403-37
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Uveitis, Intermediate; Macular Edema; Multiple Sclerosis
Keywords: Uveitis; Macular Edema; Interferon; Multiple Sclerosis; Encephalomyelitis disseminata (ED)
MeSH Terms: conditions — Uveitis, Intermediate; Macular Edema; Multiple Sclerosis; Uveitis | interventions — Interferon-beta; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interferon beta 3x weekly
  Interventions: Drug: Interferon beta
- 2 (Active Comparator): Methotrexate sc 20 mg weekly
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Interferon beta
  Arms: 1
Drug: Methotrexate
  Arms: 2

SUMMARY:
The purpose of this study is to investigate if interferon beta is superior to the standard treatment with Methotrexate for the treatment of intermediate uveitis and macular edema.

DETAILED DESCRIPTION:
Deuter et al were the first to show the anti-edematous effect of interferon alpha on inflammatory macular edema (Deuter C. M. E., Kötter I., Günaydin I., Zierhut M. Treatment of the Cystoid Macular Oedema in Behçet's Disease with Interferon Alfa-2a, Retina, in press). In an interventional, multi-centric pilot-study we could demonstrate a positive effect of interferon beta on ED associated uveitis, especially in reducing the macular edema. Undesired effects of the treatment were not observed.

Thus we want to test the efficacy and safety of interferon beta compared to standard treatment with methotrexate in a prospective, clinically controlled trial on patients who suffer from intermediate uveitis with inflammatory macular edema who either have associated ED or have no systemic disease association, i.e. primary uveitis. .

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 and over
* Active uni- or bilateral non-infectious intermediate uveitis of at least 1 year duration
* Visual acuity on the worse eye at least 0.1 (20/200) and maximally 0.6 (20/30) caused by macular edema, defined by foveal thickness ≥ 250 µm
* Either primary uveitis or diagnosis of Multiple Sclerosis
* Previous treatment with oral corticosteroids in a dose of 0.5 mg per kg bodyweight of prednisone equivalent without sufficient success
* Previous treatment with other immunosuppressive drugs is facultative

Exclusion Criteria:

* Exclusively anterior uveitis
* Absence of macular edema
* Optic nerve atrophy after neuritis nervi optici
* Peri-or intraocular injection of corticosteroids in the previous 3 months
* Allergies against any interferon
* Depression diagnosed by a psychiatrist
* Hepatic disease
* Infectious Uveitis
* Other auto-immune diseases but MS
* Pregnancy, Lactation
* Lack of reliable contraception
* Patients with metabolic, psychiatric or neoplastic diseases
* Active diseases like asthma, psoriasis or inflammatory bowel disease who have to be treated with corticosteroids
* primary or secondary immune deficiency
* Tuberculosis or other infectious lung diseases
* Hepatitis B or C
* Life vaccination during the trial duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity (3 lines ETDRS)at month 1,3,6 and 12 | at month 1,3,6 and 12

SECONDARY OUTCOMES:
Reduction of macular edema (OCT) | at month 1,3,6 and 12
Reduction intraocular inflammation (2 step change, SUN classification) | at month 1,3,6 and 12
Increase in retinal light sensitivity (fundus controlled perimetry) | at month 1,3 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Matthias D Becker, MD, PhD,FEBO, Principal Investigator — Interdisciplinary Uveitis Center, University of Heidelberg; Friederike Mackensen, MD, FEBO, Principal Investigator — Interdisciplinary Uveitis Center,University of Heidelberg; Regina Max, MD, Study Director — Interdisciplinary Uveitis Center,University of Heidelberg
Locations (1):
- Interdisciplinary Uveitis Center, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Becker MD, Heiligenhaus A, Hudde T, Storch-Hagenlocher B, Wildemann B, Barisani-Asenbauer T, Thimm C, Stubiger N, Trieschmann M, Fiehn C. Interferon as a treatment for uveitis associated with multiple sclerosis. Br J Ophthalmol. 2005 Oct;89(10):1254-7. doi: 10.1136/bjo.2004.061119. PMID 16170111